CLINICAL TRIAL: NCT01880541
Title: Assessment of Cognitive Function After Surgery in Two Types of Anesthesia (General Anesthesia Hypnosedation or Traditional) in Patients Operated for Breast Cancer
Brief Title: Assessment of Cognitive Function After Surgery in Two Types of Anesthesia in Patients Operated for Breast Cancer
Acronym: HYPNOSEIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB2009-71
Record Dates: First submitted 2012-11-06; First posted 2013-06-19 (Estimated); Results first posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-12

CONDITIONS: Patients With Breast Cancer and Breast Surgery Requiring
Keywords: Patients with breast cancer and breast surgery requiring
MeSH Terms: interventions — Hypnosis, Anesthetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypnosedation (Experimental): hypnosedation
  Interventions: Other: hypnosedation
- general anesthesia (Other): general anesthesia
  Interventions: Other: general anesthésia

INTERVENTIONS:
Other: hypnosedation — hypnosedation
  Arms: hypnosedation
Other: general anesthésia — general anesthesia
  Arms: general anesthesia

SUMMARY:
The emergence of cognitive disorders after surgery under general anesthesia (GA) is the second leading cause of patient complaints (after dental debris caused by intubation techniques). These cognitive disorders can range from simple reversible confusion (26%) with postoperative cognitive dysfunction without actual recovery (10%).

The hypnosedation is an ancient technique of anesthesia expanding its effects on cognitive function remain to this day unknown, but appear promising.

DETAILED DESCRIPTION:
For twenty years, hypnosedation is offered to patients who underwent surgery as an alternative to other anesthetic techniques (general anesthesia and locoregional), in some European and Anglo-Saxon hospitals for specific surgical indications (surgery area). It is commonly used in some hospitals.

The hypnosedation is little used in oncology

The hypnosedation is a hypnosis technique suitable for anesthesia, namely the one associated with intravenous conscious sedation and local anesthesia hypnosis. This derived from medical hypnosis Ericksoniene technique is divided into three stages:

1. induction
2. Deepening trance
3. Déhypnotisation.

This technique is currently being validated and used at national and international level, in fact it is based on 500 references and appears in the national nomenclature of the Common Classification of Medical Procedures in the code ANRP 001, states: hypnosis referred to analgesic.

ELIGIBILITY:
Inclusion Criteria:

* Female, over 18 and under 80 years
* Diagnosis of breast cancer established (Pathology)
* Life expectancy greater than 6 months
* Surgery of breast lumpectomy with or without lymph node dissection, mastectomy with or without lymph node dissection, dissection isolated
* ASA 1 (healthy patient) or 2 (patient with moderate to high function) according to the classification of the American Society of Anesthesiologist,
* Affiliation to a social security scheme,
* Information on the study, signed informed consent

Exclusion Criteria:

* Presence of major psychiatric disorders or psychotic behavior addiction, evaluated by neuropsychologist at the first preoperative consultation, through the test MINI (MINI> 4 positive responses for each module)
* Presence of neurological disorders known untreated or evaluated by neuropsychologist at the first preoperative consultation, with the MMSE test (MMSE <24)
* Patient treated morphine orally for 3 months or more
* Patient is pregnant or nursing, or of childbearing potential and not using adequate contraception,
* Patient included in another clinical study
* Inability to undergo medical monitoring study for geographical, social or psychological
* Patient deprived of liberty and most subject to a measure of legal protection or unable to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2016-11 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: COLOMBANI Sylvie, MD, Study Chair — Institut Bergonié
Locations (3):
- France (3):
  - Centre Paul Strauss, Strasbourg, Alsace
  - Institut Bergonié, Bordeaux, Aquitaine
  - Centre Oscar Lambret, Lille, Nord

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypnosedation | General Anesthesia
Started | 10 | 20
Completed | 10 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypnosedation | General Anesthesia | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (16.1) | 57.2 (11.4) | 54.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 30
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 10 | 20 | 30

OUTCOME MEASURES:

1. Primary Outcome: Presence of Cognitive Impairment
Description: Cognitive impairment is assessed using the MMSE questionnaire (MINI-MENTAL STATE EXAMINATION). the MMSE total score ranges from 0 (alteration of cognition) to 30 (no alteration)
Time Frame: on the 7th day following surgery
Population: Participants who completed the questionnaire
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hypnosedation | General Anesthesia
Number analyzed (Participants) | 10 | 19
score on a scale | 29.5 [29 to 30] | 29 [29 to 30]

2. Secondary Outcome: Presence of Cognitive Impairment
Description: Cognitive impairment is assessed using the MMSE questionnaire (MINI-MENTAL STATE EXAMINATION) The MMSE total score ranges from 0 (alteration of cognition) to 30 (no alteration)
Time Frame: 1 month after surgery
Population: Participants who completed the questionnaire
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hypnosedation | General Anesthesia
Number analyzed (Participants) | 10 | 18
score on a scale | 29.5 [29 to 30] | 30 [29 to 30]

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were not collected.
Description: Adverse events and serious adverse events were not collected.
Arm/Group | Hypnosedation | General Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2009-11-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT01880541/Prot_000.pdf